CLINICAL TRIAL: NCT06417567
Title: The Safety and Effectiveness of NEPA in Preventing Postoperative Nausea and Vomiting After General Anesthesia Gastrointestinal Cancer Surgery: A Single-Center Retrospective Study
Status: Recruiting | Type: Observational
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NEPA
Record Dates: First submitted 2024-05-12; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: General Anesthesia Gastrointestinal Cancer Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- experimental group
  Interventions: Drug: NEPA

INTERVENTIONS:
Drug: NEPA — NEPA in Preventing Postoperative Nausea and Vomiting after General Anesthesia Gastrointestinal Cancer Surgery

SUMMARY:
The rapid progress of multiple antiemetic regimens ensures that patients can receive full dose chemotherapy, however, there are still a large number of unmet clinical needs in patient evaluation and treatment. Due to the fact that patients with liver, gallbladder, and pancreatic diseases undergoing surgery are still in the stage of nausea and vomiting, the actual incidence of delayed nausea and vomiting may be underestimated. The long-term effective control of nausea and vomiting by Nitopitan Palonosetron capsules may improve the quality of life of patients during and after treatment, and ultimately improve clinical outcomes

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female, aged 18-65 years old; 2. The subjects were diagnosed with liver, gallbladder, and pancreatic diseases through histology or cytology and underwent elective surgical treatment, including but not limited to pancreaticoduodenectomy, liver resection, bile duct stone removal, etc., and received treatment with Netopitam Palonosetron capsules; 3. The subject is not in lactation period; 4. When screening female patients with potential pregnancy, it is necessary to confirm that the pregnancy test must be negative; 5. The subjects voluntarily and strictly comply with the research protocol requirements and sign a written informed consent form.

Exclusion Criteria:

* 1) Serious liver and kidney dysfunction, cardiopulmonary dysfunction, or other serious diseases have not received standardized treatment; 2) Having a serious mental illness in the past; 3) Take antiemetics or antidepressants within 48 hours before surgery; 4) Patients receiving systemic glucocorticoid treatment within 4 weeks prior to surgery; 5) Take NK1 receptor antagonists or any investigational drugs within 4 weeks prior to the start of the experiment; 6) Use CYP3A4 inducer within 4 weeks prior to surgery, and CYP3A4 substrate or potent, moderate CYP3A4 inhibitor within 1 week; 7) Pregnant or lactating women, patients with fertility who are unwilling or unable to take effective contraceptive measures; 8) Drug and/or alcohol abuse; 9) Hypocalcemia or any other condition that may cause vomiting; 10) The subject has an allergic reaction to Netopitam Palonosetron capsules or any of their excipients; 11) Participate in another clinical study within 30 days prior to baseline visit, using any exploratory drugs or devices; Allow participation in observational research; 12) Researchers assess other situations that may affect the progress of clinical research and the determination of research results.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study is a retrospective study to evaluate the efficacy and safety of Netopitam Palonosetron Capsules in preventing nausea and vomiting caused by surgical treatment in patients with liver, gallbladder, and pancreatic diseases, providing evidence-based evidence and medication basis for the use of Netopitam Palonosetron Capsules in clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete response rate within 24 hours after surgery | 3month
  defined as no vomiting, no use of rescue medication, VAS nausea score<4

SECONDARY OUTCOMES:
Complete response rates in the early postoperative period (0-2 hours), delayed period (2-24 hours), and extended observation period (24-48 hours) | Complete response rates in the early postoperative period (0-2 hours), delayed period (2-24 hours), and extended observation period (24-48 hours)
  Complete response rates in the early postoperative period (0-2 hours), delayed period (2-24 hours), and extended observation period (24-48 hours)

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No